CLINICAL TRIAL: NCT00459134
Title: A Randomized Study to Determine Whether ArginMax Improves the Sexual Function and Quality of Life in Female Cancer Survivors
Brief Title: L-Arginine Supplements in Treating Women Who Are Cancer Survivors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: IRB00001487; U10CA081851 (NIH); REBACCCWFU 97106 (Other: NCI)
Record Dates: First submitted 2007-04-09; First posted 2007-04-11 (Estimated); Results first posted 2015-01-19 (Estimated); Last update posted 2021-09-28 (Actual); Status verified 2021-09

CONDITIONS: Sexual Dysfunction; Sexuality and Reproductive Issues; Unspecified Adult Solid Tumor, Protocol Specific
Keywords: sexual dysfunction; sexuality and reproductive issues; unspecified adult solid tumor, protocol specific
MeSH Terms: conditions — Sexual Dysfunction, Physiological; Sexuality | interventions — ArginMax; Arginine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm I: ArginMax (Experimental): ArginMax® 3 pills twice daily
  Interventions: Dietary Supplement: ArginMax
- Arm II: Placebo (Placebo Comparator): Patients receive oral placebo 3 pills twice daily
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: ArginMax — Given orally
  Other Names: L-arginine
  Arms: Arm I: ArginMax
Dietary Supplement: Placebo — Given orally
  Arms: Arm II: Placebo

SUMMARY:
RATIONALE: L-arginine supplements may improve the quality of life and sexual function in women who are cancer survivors.

PURPOSE: This randomized clinical trial is studying an L-arginine supplement to see how well it works compared with a placebo in treating women who are cancer survivors.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine whether an L-arginine-based nutritional supplement (ArginMax®) improves the quality of life and sexual function in female cancer survivors.

Secondary

* Compare quality of life of patients treated with ArginMax® vs placebo.
* Compare toxicity of these regimens in these patients.
* Describe the sexual function symptom clusters (if any) in these patients.

OUTLINE: This is a randomized, double-blind, parallel-group, placebo-controlled, multicenter study. Patients are stratified according to ECOG performance status (0 or 1 vs 2 or 3), type of malignancy (pelvic vs nonpelvic), and ovarian functional status (yes vs no). Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients receive an oral L-arginine-based nutritional supplement (ArginMax®) twice daily.
* Arm II: Patients receive oral placebo twice daily. In both arms, treatment continues for 12 weeks in the absence of unacceptable toxicity.

Sexual function, quality of life, and toxicity are assessed at baseline and every 4 weeks for 12 weeks.

PROJECTED ACCRUAL: A total of 186 patients will be accrued for this study.

ELIGIBILITY:
INCLUSION CRITERIA:

Any female cancer survivor who identifies herself as concerned with her sexual quality of life and answering yes to all three of the screening questions.

* Must express interest in sexual activity
* At least 6 months following completion of all cancer therapy. Hormonal therapy and treatment with Herceptin are allowed.
* No evidence of active cancer based on physical exam and/or radiographic images obtained within 3 months of study.
* Absence of any mental, medical or physical disorder know to affect sexual function.
* No participation in another study with an investigational study drug or device during the 30 days prior to start of study drug.
* Lab values must meet the following criteria at study entry: WBC ≥ 2000, Hgb ≥ 10gm/dl, creatinine ≤ 1.5 x ULN, plt ≥ 100,000, T Bili ≤ 1.5
* ECOG performance status must be 0-2.
* Must be able to take oral medication
* Must be 18 years old or older
* Must be minority (non-white) female.

EXCLUSION CRITERIA:

* History of allergic reactions attributed to compounds of similar chemical or biologic composition to ArginMax.
* Currently taking any blood thinner such as aspirin (one 81mg aspirin, or one baby aspirin per day allowed), Persantine, Heparin, Lovenox, or Coumadin (low dose Coumadin for catheter patency is allowed).
* Patients currently taking Ginkgo Biloba are not allowed on this study.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac, arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements and/or ability for sexual function.
* Pregnant women are excluded from this study because ArginMax may be an agent with the potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with ArginMax, breastfeeding should be discontinued if the mother is treated with ArginMax.
* Because patients with immune deficiency are at increased risk of lethal infections when treated with marrow-suppressive therapy, HIV-positive patients receiving combination anti-retroviral therapy are excluded from the study because of possible pharmacokinetic interactions with ArginMax. Appropriate studies will be undertaken in patients receiving combination anti-retroviral therapy when indicated.
* Any planned surgery during study participation.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 186 (Actual)
Dates: Start 2007-05-01 (Actual); Primary Completion 2010-06-01 (Actual); Study Completion 2010-06-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kathryn M. Greven, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (25):
- United States (25):
  - CCOP - Christiana Care Health Services, Newark, Delaware
  - CCOP - Mount Sinai Medical Center, Miami Beach, Florida
  - MBCCOP - Medical College of Georgia Cancer Center, Augusta, Georgia
  - MBCCOP - JHS Hospital of Cook County, Chicago, Illinois
  - CCOP - Central Illinois, Decatur, Illinois
  - CCOP - Northern Indiana CR Consortium, South Bend, Indiana
  - Cedar Rapids Oncology Associates, Cedar Rapids, Iowa
  - MBCCOP - LSU Health Sciences Center, New Orleans, Louisiana
  - Feist-Weiller Cancer Center at Louisiana State University Health Sciences, Shreveport, Louisiana
  - CCOP - Michigan Cancer Research Consortium, Ann Arbor, Michigan
  - CCOP - Beaumont, Royal Oak, Michigan
  - CCOP - Cancer Research for the Ozarks, Springfield, Missouri
  - CCOP - Heartland Research Consortium, St Louis, Missouri
  - CCOP - St. Louis-Cape Girardeau, St Louis, Missouri
  - Hematology Oncology Associates of Central New York, PC - Northeast Center, East Syracuse, New York
  - CCOP - North Shore University Hospital, Manhasset, New York
  - Alamance Cancer Center at Alamance Regional Medical Center, Burlington, North Carolina
  - Hugh Chatham Memorial Hospital, Elkin, North Carolina
  - Southeastern Medical Oncology Center - Goldsboro, Goldsboro, North Carolina
  - Caldwell Memorial Hospital, Lenoir, North Carolina
  - Wake Forest University Comprehensive Cancer Center, Winston-Salem, North Carolina
  - CCOP - Columbus, Columbus, Ohio
  - CCOP - Main Line Health, Wynnewood, Pennsylvania
  - CCOP - Upstate Carolina, Spartanburg, South Carolina
  - CCOP - Sioux Community Cancer Consortium, Sioux Falls, South Dakota

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Arm I: ArginMax | Arm II: Placebo
Started | 94 | 92
Completed | 71 | 67
Not Completed | 23 | 25
Not completed — Physician Decision | 1 | 1
Not completed — Withdrawal by Subject | 8 | 7
Not completed — Lost to Follow-up | 6 | 7
Not completed — Surgery | 1 | 2
Not completed — Toxicity | 4 | 5
Not completed — Progression | 1 | 0
Not completed — Multiple Reasons | 2 | 3

BASELINE CHARACTERISTICS:
Population: All randomized participants
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm I: ArginMax | Arm II: Placebo | Total
Number analyzed (Participants) | 94 | 92 | 186
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 86 | 83 | 169
  >=65 years | 8 | 9 | 17
Age, Continuous [Median (Full Range); unit: years] | 51 [28 to 72] | 49 [23 to 71] | 50 [23 to 72]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 94 | 92 | 186
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 5 | 6
  Not Hispanic or Latino | 92 | 84 | 176
  Unknown or Not Reported | 1 | 3 | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 20 | 18 | 38
  White | 73 | 73 | 146
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 94 | 92 | 186

OUTCOME MEASURES:

1. Primary Outcome: Sexual Function
Description: Patients filled out the Female Sexual Function Index (FSFI) at baseline and at 4, 8, and 12 weeks following randomization. The FSFI is comprised of 2 questions related to desire, 4 questions related to arousal, 4 questions related to lubrication, 3 questions related to orgasm, 3 questions related to satisfaction, and 3 questions related to pain. Subscale scores range from 1.2 to 6 (desire) or 0 to 6 (arousal, lubrication, orgasm, and pain) or 0.8 to 6 (satisfaction). A total FSFI score is computed as the sum of the individual subscales; the overall score ranges from 2 to 36. Higher scores indicate better sexual function. The primary outcome comparison is at 12 weeks.
Time Frame: 12 weeks
Population: Participants who filled out the FSFI at any time
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Arm I: ArginMax | Arm II: Placebo
Number analyzed (Participants) | 93 | 90
units on a scale | 17.81 (0.90) | 17.15 (0.91)
Statistical Analysis 1: Comparison: Arm I: ArginMax vs Arm II: Placebo; The null hypothesis is that sexual function will be the same in both groups at 12 weeks. A Mixed effect repeated measures model constrained such that the baseline means were equal in the two groups was used to test this hypothesis; Test type: Superiority or Other; p = 0.576, Mixed Models Analysis — This p-value is not adjusted for multiple comparisons; Mixed effect repeated measures model constrained such that the baseline means were equal in the two groups; Mean Difference (Final Values) = 0.66, 95% CI 2-sided [-1.67 to 3.00], Standard Error of Mean 1.19

2. Secondary Outcome: Quality of Life
Description: Patients filled out the FACT-G quality of life questionnaire at baseline and at 4, 8, and 12 weeks following randomization. The FACT-G questionnaire is comprised of 7 questions related to physical well-being, 7 questions related to social well-being, 6 questions related to emotional well-being, and 7 questions related to functional well-being. Subscale scores range from 0 to 24 (Emotional) or 0 to 28 (Functional, Social, and Physical). A total FACT-G score is computed as the sum of the individual subscales; the overall score ranges from 0 to 108. Higher scores indicate better quality of life. The primary comparison was at 12 weeks.
Time Frame: 12 weeks
Population: Participants who filled out the FACT-G at any time
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Arm I: ArginMax | Arm II: Placebo
Number analyzed (Participants) | 93 | 92
units on a scale | 89.96 (1.38) | 85.47 (1.39)
Statistical Analysis 1: Comparison: Arm I: ArginMax vs Arm II: Placebo; The null hypothesis was that quality of life would be the same in both groups at 12 weeks. A mixed effect repeated measures model constrained such that the baseline means were equal in the two groups was used to test this hypothesis; Test type: Superiority or Other; p = 0.010, Mixed Models Analysis — This p-value is not adjusted for multiple comparisons; Mixed effect repeated measures model constrained such that the baseline means were equal in the two groups; Mean Difference (Final Values) = 4.49, 95% CI 2-sided [1.09 to 7.89], Standard Error of Mean 1.73

ADVERSE EVENTS:
Time Frame: 12 weeks
Description: The sample size for this section is the number of participants who had post-randomization toxicity data.
Arm/Group | Arm I: ArginMax | Arm II: Placebo
Serious Adverse Events (participants affected / at risk) | 6/79 | 4/77
Other Adverse Events (participants affected / at risk) | 64/79 | 60/77
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I: ArginMax (N=79) | Arm II: Placebo (N=77)
Hyperglycemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 1 (1) | 0 (0)
Hot Flashes (General disorders) | 3 (6) | 3 (4)
Infection - Vulva (Infections and infestations) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 1 (1) | 0 (0)
Pain - Abdomen (Gastrointestinal disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I: ArginMax (N=79) | Arm II: Placebo (N=77)
Headache (General disorders) | 20 (28) | 25 (46)
Hot Flashes (General disorders) | 56 (128) | 43 (107)
Nausea (Gastrointestinal disorders) | 5 (6) | 8 (11)
Neuropathy (Nervous system disorders) | 19 (38) | 11 (27)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes